CLINICAL TRIAL: NCT03800043
Title: Social Impact of Children's Dental Appearance
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Claudia Tschammler, Dr. Claudia Tschammler, Principal Investigator, University of Göttingen
Other Study IDs: 25/2/18
Record Dates: First submitted 2019-01-08; First posted 2019-01-10 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Dental Caries in Children
Keywords: Early Childhood Caries; children; dentistry; face perception; dental appearance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with own caries experience: Children with own caries experience (visible on a photo; teeth clearly visible), sufficient compliance
- Children without own caries experience: Children without own caries experience (visible on a photo; teeth clearly visible), sufficient compliance

SUMMARY:
This study evaluates the social impact of children's dental perception from children with or without caries experience. For this, children and their parents are shown pictures of child faces with healthy teeth, decayed teeth and teeth after dental treatment.

DETAILED DESCRIPTION:
Appearance and abnormalities in the face influences the life of children: attractive children get estimated as more competent and find friends easier than those with a less attractive appearance. Therefore this study aimes to evaluate the social impact of children's dental perception from children with or without own caries experience (and their parents). Both groups (with/without caries experience) are shown pictures of children with different dental status (healthy teeth, decayed teeth and teeth after dental treatment) and asked to complete established questionnaires.The division into the groups is based on photos of the children with visible teeth.

The results should be evaluated descriptively and graphically. Also the comparison between the answers of both groups for the three different dental status is planned.

ELIGIBILITY:
Inclusion Criteria:

* (parent of an child of) age 4-9 years
* sufficient compliance
* dividable into the two groups (with or without caries experience)

Exclusion Criteria:

* missing agreement to participate in the study
* insufficient compliance

Ages: 4 Years to 9 Years | Sex: All
Age Groups: Child
Study Population: children with or without caries experience and their parents
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Children: Evaluation of the whole photos | 2-3 minutes
  Questionnaire: "How would you feel having a friend looking like this?" (showing the photos of the three different dental status) (4 point face scale of Soares et al. 2015)
Children: Evaluation of the mouth on the photo | 2-3 minutes
  Questionnaire: "How would you feel having a friend with a mouth looking like this" (showing the photos of the three different dental status) (4 point face scale of Soares et al. 2015)
Children: Evaluation of their own teeth | 1-2 minutes
  Questionnaire: "How do you feel when thinking about your own teeth?" (4 point face scale of Soares et al. 2015)
Why do you feel like this? | 1-2 minutes

SECONDARY OUTCOMES:
Related parents: Evaluation of the whole photos | 1-2 minutes
  Questionnaire: Evaluate the pictures with the adjectives: clever, rude, kind, honest, confident, careful, helpful, stupid, naughty (4 point scale. 'strongly agree' = 4; 'agree' = 3; 'disagree' = 2; 'strongly disagree' = 1)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr., Study Director — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Locations (1):
- Department of Preventive Dentistry, Periodontology and Cariology, University Medical Center Goettingen, Germany, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided